CLINICAL TRIAL: NCT05783154
Title: Effect of Autologous Adipose Tissue-derived Mesenchymal Stem Cells (AT-MSCs) Therapy in Cartilage Regeneration Among Individuals With Primary Knee Osteoarthritis: A Randomized Clinical Trial
Brief Title: Effect of Mesenchymal Stem Cells in Primary Knee Osteoarthritis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Moshiur Rahman Khasru, Associate Professor, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BSMMU/2022/8897
Record Dates: First submitted 2023-02-03; First posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Osteoarthritis Knee
Keywords: Osteoarthritis; Pain; Mesenchymal Stem Cell Therapy; Physical function; Outcome, Effectiveness; Disability; Quality of Life
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Group-1) (No Intervention): In control group: 42 patients with primary KOA will receive standard conventional care including rehabilitation for knee osteoarthritis.
- Experimental Group (Group-2) (Experimental): In the interventional group, another 42 patients with primary KOA will receive adipose tissue-derived mesenchymal stem cells (AT-MSCs) injection intra-articularly (Group-2). However, group-2 (Interventional group) will be subdivided into two sub-groups namely group-2a, and group-2b. A total of 21 Participants of group-2a will receive single doses of autologous adipose tissue-derived stem cell (AT-MSCs) and standard conservative care including rehabilitation for KOA. Whereas, group-2b, 21 respondents will receive two doses of autologous adipose tissue-derived stem cell (AT-MSCs) at 3 months intervals along with standard conservative care including rehabilitation for KOA.
  Interventions: Biological: Autologous Adipose Tissue-Derived Mesenchymal Stem Cell

INTERVENTIONS:
Biological: Autologous Adipose Tissue-Derived Mesenchymal Stem Cell — After cleaning the knee with 10% povidone-iodine (Povidep10% solution, manufactured by Jayson Pharmaceuticals limited, Bangladesh) and draping it in a sterile manner, the injection site will be anesthetized with 0.5% bupivacaine (Inj. Bupi Heavy 0.5%, Manufactured by Popular Pharmaceuticals limited, Bangladesh) superficially outside of joint capsule.
  Within one hour of preparation, the autologous AT-MSC will be injected into each knee joint through medial tibio-femoral compartment in group -I using a 38-mm 18- gauge needle
  Arms: Experimental Group (Group-2)

SUMMARY:
Osteoarthritis (OA) is the most prevalent chronic joint disorder worldwide and is associated with significant pain and disability. Incidence and prevalence of osteoarthritis rise with increasing age. The prevalence of OA knee in Bangladesh seems to be higher due to poor working conditions, heavy physical labor, and occupational injuries which increase in the future. This will ultimately create a higher clinical and socioeconomic burden on the population and national economy. The course of the disease varies but is often progressive. OA of the knee is one of the common self-reported musculoskeletal pain conditions causing patients to visit the Physical Medicine and Rehabilitation (PM&R) department, at BSMMU. The primary objectives of knee OA treatment focus on pain reduction, and joint mobility improvement, as well as the reduction of disease progression and preserving patients' independence and quality of life. Current treatments aim at alleviating these symptoms by several different methods: Non-pharmacological treatments, Pharmacological treatments, and Invasive interventions. Mesenchymal stem cells (MSCs) therapies for knee osteoarthritis are being investigated in various corners of the world. Both positive and negative findings were observed in that research. Although, the effectiveness of MSCs in KOA is not yet well known. Some studies found MSCs effective, and safe in KOA, and it has the potential to regenerate/heal degraded joint cartilage. MSCs can differentiate into cartilage tissue. Furthermore, MSCs have been shown to have paracrine anti-inflammatory and immunomodulatory effects by producing different growth factors and cytokines. This therapeutics option is under investigation to date. The objective of this trial is to find the effectiveness, safety, and dose difference of adipose tissue-derived stem cells (AT-MSCs) therapy for the treatment of knee osteoarthritis (KOA).

But in fact, there is no published data about the effectiveness of autologous adipose tissue-derived mesenchymal stem cells injection on pain, joint functioning, and femoral cartilage thickness in the management of knee osteoarthritis in Bangladesh. Henceforth, this trial will generate new knowledge about the effectiveness, safety, and appropriate dose of AT-MSCs for KOA. So this research will be helpful to generate evidence-based information for an effective treatment option for the management of KOA.

ELIGIBILITY:
Inclusion Criteria:

* Primary osteoarthritis of the target knee refractory to conventional treatment only.
* Age between 40-70 years.
* All the genders.
* Participant with knee pain who fulfill 2016 revised American College of Rheumatology (ACR) criteria for OA knee
* The Kellgren and Lawrence Grade ≥2 patients.
* Pain score >3 on Visual analog scale [VAS], (0-10 cm scale).

Exclusion Criteria:

* Previous diagnosis of poly-articular disease
* Severe mechanical extra-articular deformation (>15° varus/15° valgus)
* Systemic auto-immune rheumatic disease
* Arthroscopy or intra-articular infiltration in the last 6 months
* Chronic treatment with Immunosuppressive or anticoagulant drugs
* Corticosteroids treatment in the 3 last months
* Non-steroidal anti-inflammatory drugs therapy in the last 15 days
* Poorly controlled Diabetes mellitus, blood dyscrasias
* Septic or tubercular arthritis
* Recent trauma, fracture, and unstable knee joint

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-09-16 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in the Articular Cartilage Defect | Cartilage defect will be measure before and after treatment at the month 6 and 12.
  Cartilage defect will be evaluated by MRI Osteoarthritis Knee score (MOAKS). MOAKS will be considered to describe the cartilage defect. In MOAKS the knee is divided into 14 articular sub-regions for scoring articular cartilage and Bone Marrow Lesions (BML) [0-100%] where higher score indicates more bone-marrow-lesion and the BML grades are as follows: grade 0= none, grade 1 <33%, grade 2= 33-66% and grade 3 >66%.
Changes in Femoral Cartilage thickness | Mean femoral cartilage will be measured before and after treatment at the month 6, and12.
  Femoral cartilage thickness will be measured at the three level specifically medial condyle, lateral condyle and intercondylar notch using high frequency ultrasound (Machine Model: Chison Qbit-7, Transducer: 15 mega hertz (MHz) Linear). Mean value of the three measurement will be considered for mean femoral cartilage thickness (0-4 mm).
Changes in the Pain Intensity | Pain intensity will be measured before and after treatment at the month 1, 3, 6, and12
  Pain intensity of the knee joint will be evaluated by visual analogue scale (VAS) ranges between 0 to 10 (0-10 cm scale) where score 0 indicate 'no pain' and 10 indicates 'worst pain'.
Changes in Physical functioning | Physical functioning will be measured before and after treatment at the month 1, 3, 6, and 12
  Physical functioning will be measured by The Western Ontario and McMaster Universities Arthritis Index (WOMAC) scale. WOMAC has 17 item Physical Function measure where each item score ranges between 0 to 4, and total physical function score ranges between 0-68. The higher score indicates worse physical function of the joint examined.

SECONDARY OUTCOMES:
Any Complications arises | At the month 1, 3, 6, and 12 after treatment as well as at anytime within 12 months of the treatment (if required)
  Any immediate and late complications will be documents up to 12 months after the treatment.
  All the participants will be examined for any complications during each scheduled follow-up at the month 1, 3, 6, and 12 after treatment.
  Moreover, all the participants will be asked to communicate with the investigator team for any complication/issue arises at any time within 12 months of the treatment by dedicated mobile phone number, which will be given to all the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Moshiur Rahman Khasru, MBBS, FCPS, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided
It is yet to decide by the research team